CLINICAL TRIAL: NCT02417896
Title: Pilot Non Randomised Controlled Trial of Short Term Spironolactone Use for Prevention of Acute Kidney Injury After Cardiac Surgery
Brief Title: Short Term Spironolactone for Prevention of Acute Kidney Injury After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Magdalena Madero, M.D., Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPIRO-110313
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2013-03

CONDITIONS: Acute Kidney Injuries; Kidney Injuries, Acute; Kidney Injury, Acute; Acute Renal Injury; Acute Renal Injuries
Keywords: Acute kidney injury; Spironolactone
MeSH Terms: conditions — Acute Kidney Injury | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone (Experimental): The intervention group will receive spironolactone. The drug will be administered orally to cardiac surgical patients by a study investigator (100 mg 12-24 hrs before surgery); subsequently, three further doses of 25 mg are administered orally in the morning of postoperative days 1, 2 and 3.
  Interventions: Drug: Spironolactone
- No spironolactone (No Intervention): Cardiac surgical patients requiring cardiopulmonary bypass and aortic cross clamp, randomised not to receive spironolactone will be followed for 10 days after surgery.

INTERVENTIONS:
Drug: Spironolactone — Spironolactone is administered orally to cardiac surgical patients by a study investigator (100 mg 12-24 hrs before surgery); subsequently three further doses of 25 mg are administered orally in the morning of postoperative days 1, 2 and 3. A total 1 x 100 mg and 3 x 25 mg doses of spironolactone in the intervention group will be given. If the patient has not been extubated, spironolactone is administered nasogastrically. Oral drugs will be delayed by up to 4 hours if extubation has just occurred.
  Other Names: Aldactone; Vivitar
  Arms: Spironolactone

SUMMARY:
Our aim is to test whether short term perioperative administration of oral spironolactone could reduce incidence of postoperative acute kidney injury (AKI) in cardiac surgical patients.

DETAILED DESCRIPTION:
Adult patients (>18 years old) were eligible for the study if they were undergoing elective or emergency cardiac surgery requiring CPB and aortic cross clamp. Exclusion criteria were patients with preoperative chronic renal insufficiency (Serum creatinine >1.6 mg/dl) or on dialysis, hyperkalemia (>5.0 mEq/L), AKI detected up to 24 hours before the procedure; patients receiving contrast agents 72 hours before surgery, planned off-pump cardiac surgery, hypersensitivity, allergy or known intolerance to spironolactone and pregnancy. Patients that died during the surgical procedure or 24 hours after surgery were eliminated from the analysis, as well as patients that did not receive spironolactone during the postoperative period. Criteria for stopping spironolactone were serum potassium >5.5 mEq/L, a serum creatinine level ≥2.5 mg/dL and urine output of <0.3 ml/k/hr during 8 hours.

One day prior to the procedure, patients that met the inclusion criteria were invited to participate in the trial, signing an informed consent. Spironolactone was administered orally by a study investigator (100 mg 12-24 hrs before surgery); subsequently three further doses of 25 mg were administered orally in postoperative days 1, 2 and 3. Thus, a total 1 x 100 mg and 3 x 25 mg doses of spironolactone in the intervention group were be given. If the patient had not been extubated, spironolactone was administered nasogastrically. Oral drugs were delayed by up to 4 hours if extubation had just occurred. The patients that decided not to receive spironolactone were followed during the study period and considered as controls. Preexisting ACE inhibitor, angiotensin receptor blocker, or MR antagonist were not suspended before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Elective and emergent cardiac surgery with cardiopulmonary bypass and aortic cross clamp

Exclusion Criteria:

* Patients with preoperative chronic renal insufficiency on dialysis
* Acute kidney injury detected up to 24 hours before the procedure a
* Patients receiving contrast agents 72 hours before surgery
* Planned off-pump cardiac surgery
* Hypersensitivity, allergy or known intolerance to spironolactone
* Pregnancy
* Hyperkalemia with potassium >5.0 mEq/L

Criteria for stopping study medication:

- Serum potassium >5.5 mEq/L

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury (AKI) defined by the AKIN criteria in patients submitted to cardiac surgery with spironolactone therapy. | First 10 days after cardiac surgery

SECONDARY OUTCOMES:
Change in urinary neutrophil gelatinase-associated lipocalin (NGAL) concentration. | First 10 days after cardiac surgery
  Change in urinary neutrophil gelatinase-associated lipocalin (NGAL) concentration in patients submitted to cardiac surgery with or without previous spironolactone therapy.
Mortality | First 10 days after cardiac surgery
  Mortality in patients submitted to cardiac surgery with or without previous spironolactone therapy.
Hyperkalemia | First 10 days after cardiac surgery
  Hyperkalemia in patients submitted to cardiac surgery with or without previous spironolactone therapy.
Renal replacement therapy | First 10 days after cardiac surgery
  Renal replacement therapy in patients submitted to cardiac surgery with or without previous spironolactone therapy.
Length of stay in intensive care unit | First 20 days after cardiac surgery
  Length of stay in intensive care unit or patients submitted to cardiac surgery with or without previous spironolactone therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Gamba, PhD, Study Director — Instituto Nacional de la Nutrición Salvador Zubiran
Locations (2):
- Mexico (2):
  - Instituto Nacional de la Nutrición Salvador Zubirán, Mexico City, Mexico City
  - Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Mexico City

REFERENCES:
- [Background] Barrera-Chimal J, Perez-Villalva R, Rodriguez-Romo R, Reyna J, Uribe N, Gamba G, Bobadilla NA. Spironolactone prevents chronic kidney disease caused by ischemic acute kidney injury. Kidney Int. 2013 Jan;83(1):93-103. doi: 10.1038/ki.2012.352. Epub 2012 Sep 26. PMID 23014458
- [Background] Sanchez-Pozos K, Barrera-Chimal J, Garzon-Muvdi J, Perez-Villalva R, Rodriguez-Romo R, Cruz C, Gamba G, Bobadilla NA. Recovery from ischemic acute kidney injury by spironolactone administration. Nephrol Dial Transplant. 2012 Aug;27(8):3160-9. doi: 10.1093/ndt/gfs014. Epub 2012 Apr 19. PMID 22516623
- [Background] Barrera-Chimal J, Perez-Villalva R, Cortes-Gonzalez C, Ojeda-Cervantes M, Gamba G, Morales-Buenrostro LE, Bobadilla NA. Hsp72 is an early and sensitive biomarker to detect acute kidney injury. EMBO Mol Med. 2011 Jan;3(1):5-20. doi: 10.1002/emmm.201000105. Epub 2010 Dec 14. PMID 21204265
- [Background] Prowle JR, Calzavacca P, Licari E, Ligabo EV, Echeverri JE, Haase M, Haase-Fielitz A, Bagshaw SM, Devarajan P, Bellomo R. Pilot double-blind, randomized controlled trial of short-term atorvastatin for prevention of acute kidney injury after cardiac surgery. Nephrology (Carlton). 2012 Mar;17(3):215-24. doi: 10.1111/j.1440-1797.2011.01546.x. PMID 22117606
- [Background] Pretorius M, Murray KT, Yu C, Byrne JG, Billings FT 4th, Petracek MR, Greelish JP, Hoff SJ, Ball SK, Mishra V, Body SC, Brown NJ. Angiotensin-converting enzyme inhibition or mineralocorticoid receptor blockade do not affect prevalence of atrial fibrillation in patients undergoing cardiac surgery. Crit Care Med. 2012 Oct;40(10):2805-12. doi: 10.1097/CCM.0b013e31825b8be2. PMID 22824930
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152